CLINICAL TRIAL: NCT04234932
Title: Short-term Effect of Rho-kinase Inhibitor on Retinal Circulation
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of the Incarnate Word (Other)
Responsible Party: Principal Investigator, Richard Trevino, OD, FAAO, Principal Investigator, University of the Incarnate Word
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 19-12-005
Record Dates: First submitted 2020-01-15; First posted 2020-01-21 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Netarsudil alone (Experimental): Topical application of netarsudil 0.02%
  Interventions: Drug: Netarsudil Ophthalmic
- Netarsudil plus latanoprost (Active Comparator): Topical application of netarsudil 0.02% with latanoprost 0.005%
  Interventions: Drug: Netarsudil Ophthalmic

INTERVENTIONS:
Drug: Netarsudil Ophthalmic — Topical instillation of commercial preparations of netarsudil 0.02% ophthalmic solution (Rhopressa and Roclatan)
  Other Names: Latanoprost Ophthalmic

SUMMARY:
Investigate changes in optical coherence tomography angiography of the optic nerve and macula following topical instillation of commercial preparations of netarsudil 0.02% ophthalmic solution.

ELIGIBILITY:
Inclusion Criteria:

* Normal ocular health

Exclusion Criteria:

* Females who are or may be pregnant or who are nursing
* Uncontrolled hypertension
* Allergy to netarsudil or latanoprost

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Peripapillary capillary perfusion density | 90 minutes
  Mean change in peripapillary capillary perfusion as assessed using optical coherence tomography angiography

SECONDARY OUTCOMES:
Macular capillary perfusion density | 90 minutes
  Mean change in macular capillary perfusion as assessed using optical coherence tomography angiography

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Incarnate Word, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared